CLINICAL TRIAL: NCT02923323
Title: Cross-sectional, Case Control Study of Electrical Activity and Neurocognitive Performance During Hyperglycemia and Near Normoglycemia, and Brain Tissue Integrity in Children and Youth With Type 1 Diabetes and in Healthy Population
Brief Title: Neurocognitive Performance During Hyperglycemia , and Brain Tissue Integrity in Youth With Type 1 Diabetes and in Healthy
Acronym: T1DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Bar-Ilan University, Israel (Other); Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Marianna Rachmiel, Dr. Marianna Rachmiel, Assaf-Harofeh Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 97/14
Record Dates: First submitted 2015-07-08; First posted 2016-10-04 (Estimated); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Neurocognitive Function; MRI; Diffusion Tensor Imaging (DTI); Sleep
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Electroencephalography; Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 T1DM aged 12-18 years. (Experimental): T1DM patients. Receiving regularly insulin. Interventions: performance of continuous EEG , CGMS, MRI of brain with DTI , actigraph, neurocognitive testing
  Interventions: Device: MRI including DTI , EEG, CGMS; Behavioral: Neurocognitive tests
- Group 2 Healthy aged 12-18 years. (Active Comparator): Healthy Interventions: performance of continuous EEG , CGMS, MRI of brain with DTI , actigraph, neurocognitive testing
  Interventions: Device: MRI including DTI , EEG, CGMS; Behavioral: Neurocognitive tests

INTERVENTIONS:
Device: MRI including DTI , EEG, CGMS — Will be connected to continuous simultaneous systems
Behavioral: Neurocognitive tests — Will perform multiple tests of neurocognitive functions after lunch

SUMMARY:
Study population : 90 Participants. 60 with T1DM , and 30 healthy controls. T1DM patients will be recruited by research publication in diabetes mellitus forums.

Baseline visit: informed consent signing. Medical history data, vital signs, physical exam and neurocognitive testing. Capillary glucose prior to testing > 70 mg/dl.

Session 2 - combined simultaneous EEG , continuous glucose monitor system (CGMS) assessment, neurocognitive testing, and sleep quality assessment.

Participants will be hospitalized for 30 hours in the continuous-EEG unit at the Pediatric Neurology Department, Assaf-Harofeh Medical Center. Continuous simultaneous EEG and CGMS monitoring, and two separate sessions of neurocognitive assessments at glucose > 240 mg/dl and at glucose < 180 mg/dl, respectively.

Neurocognitive assessment will be performed after lunch on day 1, and after lunch on day 2. Day 1, regular insulin dose before lunch, and a cognitive assessment which will be performed with glucose level > 70 mg/dl and below 180 mg/dl.

On day 2, with no regular insulin dose before lunch and the same cognitive test will be performed with glucose level > 240 mg/dl During the 30 hours the participants will be connected to continuous EEG recording, sleep monitoring and CGMS. The study participants and research team will be blinded to the EEG and CGMS readings while recorded.

Participants will be able to convey their daily activities in their room. They will have their regular diet and regular daily activities.

Participants will measure at least 4 blood glucose measurements by prick tests, insulin management by multiple daily injections or pump therapy and meals.

Healthy participants will measure twice daily as required for CGMS calibration. The participants will stay connected to the CGMS for additional 4 days at their home setting for complete sleep quality assessment by sleep diary and actigraph.

The first night in hospital is to assess the association between actigraph and EEG and CGMS variability. The 4 nights at home are for assessment of CGMS, quality of life and actigraph readings.

Control group (healthy) will perform only one session of neurocognitive studies on day 1, after lunch with no insulin injection and will be discharged after 24 hours, with the CGMS and actigraph

DETAILED DESCRIPTION:
An inter-disciplinary repeated measures case control design study is proposed, whereby novel methods of brain imaging, brain electrophysiological activity, neuropsychological tests will be examined in concert with the children's dynamic changes in glucose levels. This will be compared to healthy population.

Study population Participants with T1DM and healthy siblings will be recruited by research publication in diabetes mellitus forums, and through the Pediatric Endocrinology Association. It will include mainly participants from the Pediatric Diabetes Mellitus Clinics at Assaf Harofeh; however, every child who complies with the inclusion and exclusion criteria will be recruited.

Inclusion criteria: Families living in areas with high access to medical care. Age: 12-18 years old having diagnosed with T1DM for longer than 2 years.

Exclusions: head injuries, epileptic episodes, psychiatric medications, lack of Hebrew abilities, disagreement to keep with all study requests, history of more than one episode of severe hypoglycemic event in the past, including loss of consciousness or more than one episode of diabetic ketoacidosis (DKA) . Patients with significant renal or liver function abnormalities will be excluded.

Similar exclusion criteria for healthy control population. All parents will sign informed consent and children will assent, according to Ethics committee regulations, prior to beginning study sessions.

Procedures:

Study design includes 3 sessions, which will be performed during a period of 2 -12 weeks, according to participants' convenience.

The data acquired in each session will be analyzed both within groups and among groups in order to evaluate possible descriptive variables to performance differences among diabetic patients in addition to the expected differences between healthy and diabetic adolescents, and the expected difference between T1DM patients with variable glycemic control.

Session 1 - baseline visit:

Signing parents' informed consent and participant assent. Medical history intake by the study physician including physical exam. Data regarding age of diagnosis, DKA at diagnosis, history of serious hypoglycemic or DKA events, management profile, annual average HbA1c, systems review, chronic medical diseases, medications will be provided from parents, patients and summary letters and from clinical care charts.

Physical examination will be performed including blood pressure, pulse, weight, height, BMI, pubertal stage, injection sites.

Specialized psychological neurocognitive team will perform neurocognitive studies to one of the parents and participants. Tests will be performed in a clinic setting in order to provide a baseline cognitive and lingual ability to continue in the next study sessions. Capillary glucose assessment will be performed prior to testing to ensure glucose > 70 mg/dl.

The neurocognitive studies will include an extensive battery of cognitive assessments, including tasks that were specifically designed for the purposes of the current project [Estimation Time task, Continuous Performance Test (CPT), Emotional Stroop for eating disorders (EST-ED) and New objects memory task]. Tasks will be performed in part by computer provided tasks and partly by hand written tasks.

Session 2 - combined simultaneous EEG and CGMS assessment visit, and sleep quality assessment:

Participants will be hospitalized for 30 hours in the continuous-EEG unit at the Pediatric Neurology Department, Assaf-Harofeh Medical Center, where they will undergo 30 hr. continuous simultaneous EEG and CGMS monitoring, and two separate sessions of neurocognitive assessments at glucose > 240 mg/dl and at glucose < 180 mg/dl, respectively.

They will arrive to the EEG unit after breakfast on day 1. They will be connected to both systems and accuracy assessment will be performed before lunchtime of day 1. They will remain in unit, attached to both systems until afternoon on day 2, a total of 30 hours.

Neurocognitive assessment will be performed after lunch on day 1, and after lunch on day 2.

On day 1, they will receive their regular insulin dose before lunch, and a cognitive assessment which will be performed with glucose level > 70 mg/dl and below 180 mg/dl.

On day 2, they will not receive their regular insulin dose before lunch, and the same cognitive test will be performed with glucose level > 240 mg/dl. An episode of food intake without a bolus of insulin occurs unfortunately very often among adolescents in daily life.

The neurocognitive assessment performed at this session will include working memory, selective attention and inhibitory control tasks: Test of Memory and Learning (TOMAL) , selective attention, cognitive flexibility and and inhibitory control (cognitive and emotional Stroop tasks) , word fluency test , visual memory and executive functions (ROCF) ; visuospatial short-term working memory ; auditory verbal learning ; Towers of Hanoi, a computerized task based on Tower of London (TOL). number storage capacity of working memory as well as tests of executive (WISC-IV) .

During the 30 hours the participants will be connected to continuous EEG recording, sleep monitoring and CGMS. The study participants and research team will be blinded to the EEG readings while recorded. The study team and participants will not be blinded to the CGMS recording.

Participants will be able to convey their daily activities in their room, while monitored by continuous EEG. They will have their regular diet and regular daily activities.

Participants will carry on with their regular daily routine of at least 4 blood glucose measurements by prick tests, insulin management by multiple daily injections or pump therapy and meals.

Participants from group 3 will measure glucose by prick test only twice daily as required for CGMS calibration.

During 5 consecutive nights, including the night in hospital, the participants will be assessed for sleep quality by sleep diary and actigraph.

The first night in hospital is to assess the association between actigraph and EEG and CGMS variability. The 4 nights at home are for assessment of CGMS, quality of life and actigraph readings.

Session 3 - brain imaging :

MRI scans including T1, T2, DTI and vascular MRI. All subjects will undergo anatomic (T1, T2) scans, DTI scans, and vascular scan. The session length will be of 20 -30 minutes max. The procedure will be performed with no sedation administration , no contrast material.

Description of measures used in the study:

Neurocognitive and psychosocial questionnaire and tasks based Continuous EEG monitoring This is a non-invasive method of examination, recording electrical cerebral brain activity (electroencephalographic reading) for continuous prolonged periods of hours and days, without causing inconvenience to the subjects. Results are of high resolution and reliability.

The patients will be connected to a standard digital acquisition EEG machine (Bio-logic Systems corp, Electro-Cap International Inc, Illinois) by 19 scalp electrodes applied according to the 10-20 system and one cardiac electrode for simultaneous electrocardiographic (ECG) assessment. The EEG acquisition will be performed at sampling rate of 256 Hz.

The EEG data from all subjects will be exported to the Matlab environment. Matlab is a computing language permitting more efficient analysis of data that are computationally intensive (The Mathworks Inc, MA).

Spectral analysis of the EEG signal will be performed by fast Fourier Transform (FFT - using MATLAB function) for each patient on 2 seconds epochs of recording, taken at 5 minutes intervals (to fit the frequency of CGMS measurements), with a resolution of 0.5 Hz. The frequency bands will be divided to delta (0.5-3.5 Hz), theta (4-7.5 Hz), alpha (8-13 Hz), beta (13.5-29.5 Hz), low gamma (30-47.5 Hz) and high gamma (52.5-80 Hz).

Each participant will have 3 electrodes connected to chest to see consecutive ECG measurements.

continuous glucose monitoring by - CGMS The CGMS (Minimed Inc., Sylmar. Calif) is a portable device allowing continuous measurements of interstitial glucose concentration (IGC) by a disposable subcutaneous catheter, operated by a cable and monitor system. The system measures glucose values every 10 seconds and stores an average value every 5 minutes, providing 288 measures per day [26]. The system reports values in the range between 40-400 mg/dl (glucose values lower than 40 mg/dl are reported as 40 mg/dl and values above 400 mg/dl are reported as 400 mg/dl). The median correlation of the device to capillary glucose is 0.92, with 75% of the correlation values above 0.75, 96.3% of the reference values in the range of >216 mg/dl are accurate. Calibration and verification of IGC will be performed prior to all meals and at bedtime, according to capillary measured glucose levels by finger taps, using a conventional glucometer. Data will be downloaded by using CGMS solutions software, transformed to Excel datasheet, and analyzed by a Pediatric Endocrinologist.

Pittsburgh Sleep Quality Index (PSQI) The PSQI is a well-validated 19-item self-report measure of sleep quality in adults over the previous month. The PSQI provides a global score of sleep quality and seven sub scale scores. A total score of ≥ 5 has been recommended as clinically significant in terms of poor sleep quality. The PSQI has demonstrated good validity and reliability (Cronbach's α > 0.8). Participants will complete the PSQI during session 2, during day 1, prior to wearing the actigraph. The questionnaire is attached in appendix 2.

Actigraphy An Actigraph (Micro-mini-Motion logger, Ambulatory Monitoring Inc., Ardsley, New York , USA) is a wrist-watch sized motion detector that has been shown to be highly valid and reliable for differentiating sleep from wakefulness, as well as recording total sleep time (r=97 compared to polysomnography). Participants will wear an actigraph for 5 consecutive nights on their nondominant wrist. Sleep patterns will be estimated using the validated Sadeh scoring algorithm developed for adolescents. Actigraph sleep measures included: (a) sleep onset/ bedtime; (b) sleep offset/wake time, (c) time in bed (minutes from sleep onset to sleep offset), (d) actual sleep time (number of sleep minutes between sleep onset and sleep offset), (e) sleep efficiency (actual sleep time divided by time in bed, expressed as a percent), (f) longest sleep period (longest consecutive period scored as sleep without any identified awakening), (g) median number of nighttime wakings (at least 5 consecutive minutes), and (h) median length of nighttime waking.

Sleep Diary During the nights participants will wear the actigraph at home, they will be asked to rate every day their previous nights' sleep using a very short questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Families living in areas with high access to medical care.
* Age:12-18 years old having diagnosed with T1DM for longer than 2 years.

Exclusion Criteria:

* Head injuries
* Epileptic episodes
* Psychiatric medications
* Lack of Hebrew abilities
* Disagreement to keep with all study requests
* History of more than one episode of severe hypoglycemic event in the past including loss of consciousness or more than one episode of diabetic ketoacidosis.
* Patients with significant renal or liver function abnormalities.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Association between interstitial glucose concentration and EEG power | 2 years
  continuous monitoring of both EEG readings and glucose

SECONDARY OUTCOMES:
Association between interstitial glucose concentration and neurocognitive functions | 2 years
  Association between glucose concentration in mg/dl and scoring on tests. The neurocognitive tests have numerical scoring. Those scores will be assessed according to glucose levels in the T1D group and health group in separate and between groups.

OTHER OUTCOMES:
association between quality of sleep and glycemic control | 2 years
  Quality of sleep will be assessed according to actigraph and correlated with HbA1c levels , and compared between groups
DTI assessment of brain MRI according to HbA1c | 2 years
  Brain DTI parameters will be compared between healthy and T1DM groups

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Rachmiel, M.D, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Haroffeh Medical center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: No